CLINICAL TRIAL: NCT06077916
Title: The Efficiency and Safety of Intravenous Azithromycin in Preparation of Endoscopy for Upper Gastrointestinal Bleeding
Brief Title: Gastric CLEANsing by Intravenous AZithromycin in Urgent Endoscopy
Acronym: CLEAN-AZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Colentina (Other)
Collaborators: Spitalul clinic judetean de urgenta Craiova (Unknown); Spitalul clinic judetean de urgenta "Pius Brinzeu", Timisoara (Unknown); Spitalul universitar de urgenta Elias, Bucuresti (Unknown); Spitalul clinic de urgenta, Bucuresti (Unknown); Spitalul clinic Judetean de Urgenta, Constanta (Unknown); Spitalul Clinic de Urgenţǎ Bucureşti (Unknown); Spitalul Universitar de Urgenta Militar Bucuresti (Unknown); Spitalul Judetean de Urgenta Tulcea (Unknown); Spitalul de Urgenta Prof. Dr. Agrippa Ionescu (Unknown); Spitalul Universitar de Urgență București (Unknown); Institutul de Gastroenterologie si Hepatologie Iasi (Unknown); Institutul Regional de Gastroenterologie si Hepatologie Prof.dr.Octavian Fodor, Cluj (Unknown)
Responsible Party: Principal Investigator, Andrei Voiosu, Investigator, Clinical Hospital Colentina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 10/27.03.2023
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Azithromycin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): iv perfusion of 250 mL of 0.9% saline solution
  Interventions: Drug: Saline solution
- Azithromycin (Experimental): iv perfusion of 500 mg azithromycin in 250 mL of 0.9% saline solution
  Interventions: Drug: Azithromycin; Drug: Saline solution

INTERVENTIONS:
Drug: Azithromycin — azithromycin is reconstituted and administered according to standard prescription indications in 250 mL saline solution
  Arms: Azithromycin
Drug: Saline solution — placebo consisting of saline solution 250 mL is administered

SUMMARY:
This study will test the hypothesis that azythromycin is efficient and safe in cleansing the upper gastrointestinal tract for endoscopic examination in the case of acute bleeding.

DETAILED DESCRIPTION:
In this study patients with upper GI bleeding will be randomzied to either i.v. azythromycin or placebo in order to evaluate the efficiency and safety of azythromycin for upper GI cleanliness during diagnostic endoscopy. A validated upper GI cleanliness score (Toronto score with values up to 10) and a visual analog scale will be used to evaluate cleanliness. Need for repeat endoscopy due to poor preparation, duration of hospitalization and requirement for blood transfusions during hospitalization will also be assessed as will any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* acute upper GI bleeding (<12 hours)

Exclusion Criteria:

* prokinetics <12 hours
* allergy to azithromycin
* use of contraindicated drugs (due to interactions)
* pregnancy
* physician option

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Toronto Upper Gastrointestinal Cleaning Score | up to 12 hours after admission
  Quality of endoscopic visualization during urgent upper GI endo according to the Toronto Score (higher scores >8/12 mean good bowel cleanliness)
Need for second look endoscopy | up to 48 hours after endoscopy
  Physician judgement on need for repeat endoscopy due to low Toronto score

SECONDARY OUTCOMES:
Toronto Upper Gastrointestinal Cleaning Score | up to 12 hours
  visualization quality per upper GI segment
Total hospitalization | one month
  total duration of hospital stay
Number of blood units transfused | one month
  Number of blood units transfused
Adverse events | one month
  all advers events
Duration of endoscopy | up to 12 hours after admission
  Duration of endoscopy
Score of endoscopist satisfaction on a 4-item scale | up to 12 hours
  semiquantitative measure of satisfaction with cleanliness of the upper GI tract according to visual analog scale of 5-items

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Mateescu, Prof, Principal Investigator — Clinical Hospital Colentina
Locations (1):
- Colentina Clinical Hospital, Bucharest, Bucharest, Romania